CLINICAL TRIAL: NCT00334802
Title: Combination Study of LY188011 and Paclitaxel in Patients With Metastatic/Recurrent Breast Cancer After Neo-adjuvant/Adjuvant Chemotherapy With Anthracycline
Brief Title: Combination Chemotherapy of Gemcitabine and Paclitaxel for Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9066; B9E-JE-MB22 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-06-06; First posted 2006-06-08 (Estimated); Results first posted 2009-07-20 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: gemcitabine; Drug: paclitaxel

INTERVENTIONS:
Drug: gemcitabine — Phase 1: 1000 mg/m2, intravenous (IV), day 1 and day 8 x 2 cycles (dose escalation)
  Phase 2: dose determined by phase 1
  Other Names: LY188011; Gemzar
Drug: paclitaxel — Phase 1: 175 mg/m2, intravenous (IV), every 21 days x 2 cycles
  Phase 2: 175 mg/m2, intravenous (IV), every 21 days x 2 cycles

SUMMARY:
To investigate efficacy, safety and PK of gemcitabine and paclitaxel combination in patients with metastatic breast cancer after adjuvant/neo-adjuvant chemotherapy with anthracycline regimen

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed breast cancer
* Received adjuvant/neo-adjuvant chemotherapy for breast cancer with anthracycline regimen
* To have at least one measurable region
* Eastern Cooperative Oncology Group (ECOG) Performance Status: 0-1
* To have adequate organ function (bone marrow, liver and renal function)

Exclusion Criteria:

* To have interstitial pneumonia or pulmonary fibrosis
* To have inflammatory breast cancer
* Within 28 days after the latest chemotherapy or radiotherapy, 14 days after the latest hormonal/immunotherapy or 7 days after surgery
* To have brain metastases with symptoms
* To have severe complication (cardiac infarction, infection, drug hypersensitivity or diabetes)

Ages: 20 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-06; Primary Completion 2008-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- Japan (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ehime
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Numakunai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Gemcitabine: 1000 mg/m2, intravenous (IV), day 1 and day 8 x 2 cycles Paclitaxcel: 175 mg/m2, intravenous (IV), every 21 days x 2 cycles
- Dose Level 2: Gemcitabine: 1250 mg/m2, intravenous (IV), day 1 and day 8 x 2 cycles Paclitaxcel: 175 mg/m2, intravenous (IV), every 21 days x 2 cycles
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2
Started | 6 | 56
Completed | 0 | 16
Not Completed | 6 | 40
Not completed — Progressive Disease | 2 | 24
Not completed — Toxicity | 1 | 5
Not completed — Lack of Efficacy | 1 | 3
Not completed — Patient Condition Aggrevated | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Adverse Event | 0 | 3
Not completed — Criteria for Starting Next Cycle Not Met | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Total
Number analyzed (Participants) | 6 | 56 | 62
Age Continuous [Mean (Standard Deviation); unit: years] | 58.2 (4.49) | 54.4 (8.73) | 54.7 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 56 | 62
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 6 | 56 | 62
Age at Primary Diagnosis [Number; unit: participants]
  <30 years old | 0 | 0 | 0
  30 to <40 years old | 0 | 3 | 3
  40 to <50 years old | 1 | 20 | 21
  50 to <60 years old | 3 | 24 | 27
  60 to <70 years old | 2 | 8 | 10
  ≥70 years old | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 4 | 50 | 54
    1 - Ambulatory, Restricted Strenuous Activity | 2 | 6 | 8
Body Weight [Mean (Standard Deviation); unit: kilograms] | 57.18 (15.313) | 55.76 (8.715) | 55.90 (9.375)
Height [Mean (Standard Deviation); unit: centimeters] | 153.53 (7.987) | 154.71 (6.184) | 154.60 (6.312)

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Best response recorded from the start of treatment until disease progression/recurrence using Response Evaluation Criteria In Solid Tumors (RECIST) criteria that defines when participants improve ("respond"), stay the same ("stable"), or worsen ("progression") during treatment. Responders are patients with complete response or partial response.
Time Frame: baseline to measured progressive disease
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 6 | 56
participants
  Complete Response | 0 | 0
  Partial Response | 3 | 25
  Stable Disease | 1 | 17
  Progressive Disease | 1 | 11
  Not Evaluable | 1 | 3
Statistical Analysis 1: Comparison: Dose Level 1; Test type: Superiority or Other; p = 0.169, t-test, 2 sided — P-value for Dose Level 1 Responders (Complete Response + Partial Response)
Statistical Analysis 2: Comparison: Dose Level 2; Test type: Superiority or Other; p = 0.001, t-test, 2 sided — P-value for Dose Level 2 Responders (Complete Response + Partial Response)

2. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of progression or death as a result of any cause.
Time Frame: time of response to progressive disease
Measure: Median (Full Range); unit: months
Arm/Group | Dose Level 2
Number analyzed (Participants) | 56
months | 4.70 [1.2 to 7.3]

3. Secondary Outcome: Time to Progressive Disease
Description: Defined as the time from study enrollment to the first date of disease progression. Time to disease progression was censored at the date of death if death was due to other cause.
Time Frame: baseline to measured progressive disease
Measure: Median (Full Range); unit: days
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 6 | 56
days | 310.5 [42 to 455] | 194.0 [29 to 265]

4. Secondary Outcome: Number of Participants Alive at One Year (1-Year Survival)
Time Frame: baseline to date of death from any cause, evaluated at 1 year
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 6 | 56
participants | 5 | 45

5. Secondary Outcome: Pharmacokinetics - Maximum Plasma Concentration (Cmax)
Description: Maximum plasma concentration of gemcitabine plus paclitaxel on Day 1, Cycle 1, and gemcitabine monotherapy on Day 8, Cycle 1.
Time Frame: cycle 1, day 1 (0 minutes, 3, 3.25, 3.5, 3.58, 3.75, 4, 4.5, 5 hours) and 8 (0, 15, 30, 35, 45, 60, 90, 120 minutes)
Population: Six participants from each dose level (Dose Level 1 and Dose Level 2) were assessed for pharmacokinetic variables.
Measure: Geometric Mean (Full Range); unit: nanograms per milliliter (ng/mL)
Groups:
- Gemcitabine + Paclitaxcel: Gemcitabine: 1000 mg/m2, intravenous (IV), day 1 and day 8 or Gemcitabine: 1250 mg/m2, intravenous (IV), day 1 and day 8 Paclitaxcel: 175 mg/m2, intravenous (IV), day 1
- Gemcitabine: Gemcitabine: 1000 mg/m2, intravenous (IV), day 1 and day 8 or Gemcitabine: 1250 mg/m2, intravenous (IV), day 1 and day 8
Arm/Group | Gemcitabine + Paclitaxcel | Gemcitabine
Number analyzed (Participants) | 12 | 12
nanograms per milliliter (ng/mL) | 25800 [12800 to 43600] | 25400 [20000 to 33100]

6. Secondary Outcome: Pharmacokinetics - Area Under the Concentration Curve (AUC)
Description: Area under the concentration curve from time zero to infinity.
Time Frame: cycle 1, day 1 (0 minutes, 3, 3.25, 3.5, 3.58, 3.75, 4, 4.5, 5 hours) and 8 (0, 15, 30, 35, 45, 60, 90, 120 minutes)
Population: Six participants from each dose level (Dose Level 1 and Dose Level 2) were assessed for pharmacokinetic variables.
Measure: Geometric Mean (Full Range); unit: nanograms*hour per milliliter (ng*hr/mL)
Arm/Group | Gemcitabine + Paclitaxcel | Gemcitabine
Number analyzed (Participants) | 12 | 12
nanograms*hour per milliliter (ng*hr/mL) | 16300 [11700 to 25500] | 14700 [11500 to 21000]

7. Secondary Outcome: Pharmacokinetics - Half Life (t½)
Description: Apparent elimination half-life.
Time Frame: cycle 1, day 1 (0 minutes, 3, 3.25, 3.5, 3.58, 3.75, 4, 4.5, 5 hours) and 8 (0, 15, 30, 35, 45, 60, 90, 120 minutes)
Population: Six participants from each dose level (Dose Level 1 and Dose Level 2) were assessed for pharmacokinetic variables.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | Gemcitabine + Paclitaxcel | Gemcitabine
Number analyzed (Participants) | 12 | 12
hours | 0.282 [0.192 to 1.00] | 0.258 [0.162 to 0.969]

ADVERSE EVENTS:
Arm/Group | Dose Level 1 | Dose Level 2
Serious Adverse Events (participants affected / at risk) | 1 | 3
Other Adverse Events (participants affected / at risk) | 6 | 56
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Dose Level 1 | Dose Level 2
Haemoglobin decreased (Investigations) | 1/6 (1) | 0/56 (0)
Pneumonia (Infections and infestations) | 0/6 (0) | 1/56 (1)
Anorexia (Metabolism and nutrition disorders) | 0/6 (0) | 1/56 (1)
Panic disorder (Psychiatric disorders) | 0/6 (0) | 1/56 (1)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Dose Level 1 | Dose Level 2
Bronchitis (Infections and infestations) | 1/6 (1) | 0/56 (0)
Cystitis (Infections and infestations) | 1/6 (1) | 2/56 (2)
Folliculitis (Infections and infestations) | 1/6 (1) | 0/56 (0)
Nasopharyngitis (Infections and infestations) | 1/6 (2) | 17/56 (26)
Tinea infection (Infections and infestations) | 1/6 (1) | 0/56 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/6 (1) | 7/56 (10)
Anorexia (Metabolism and nutrition disorders) | 3/6 (5) | 27/56 (54)
Insomnia (Psychiatric disorders) | 1/6 (1) | 13/56 (17)
Dysgeusia (Nervous system disorders) | 2/6 (5) | 19/56 (57)
Headache (Nervous system disorders) | 2/6 (5) | 15/56 (36)
Hypoaesthesia (Nervous system disorders) | 2/6 (3) | 20/56 (42)
Dizziness (Nervous system disorders) | 1/6 (1) | 5/56 (7)
Neuropathy peripheral (Nervous system disorders) | 1/6 (1) | 13/56 (18)
Sensory disturbance (Nervous system disorders) | 1/6 (1) | 13/56 (13)
Palpitations (Cardiac disorders) | 2/6 (2) | 2/56 (2)
Angiopathy (Vascular disorders) | 2/6 (3) | 25/56 (73)
Flushing (Vascular disorders) | 1/6 (1) | 5/56 (11)
Hypertension (Vascular disorders) | 1/6 (2) | 1/56 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1/6 (1) | 10/56 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1/6 (2) | 4/56 (6)
Nausea (Gastrointestinal disorders) | 3/6 (10) | 29/56 (105)
Constipation (Gastrointestinal disorders) | 1/6 (3) | 13/56 (63)
Vomiting (Gastrointestinal disorders) | 1/6 (2) | 16/56 (38)
Alopecia (Skin and subcutaneous tissue disorders) | 4/6 (4) | 34/56 (34)
Erythema (Skin and subcutaneous tissue disorders) | 2/6 (2) | 9/56 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 2/6 (2) | 10/56 (25)
Eczema (Skin and subcutaneous tissue disorders) | 1/6 (1) | 12/56 (22)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1/6 (1) | 3/56 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 1/6 (1) | 1/56 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/6 (1) | 23/56 (69)
Arthritis (Musculoskeletal and connective tissue disorders) | 1/6 (2) | 0/56 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1/6 (2) | 6/56 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 1/6 (11) | 19/56 (62)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/6 (1) | 12/56 (31)
Malaise (General disorders) | 5/6 (22) | 34/56 (116)
Oedema peripheral (General disorders) | 2/6 (4) | 6/56 (10)
Pyrexia (General disorders) | 2/6 (3) | 16/56 (47)
Chills (General disorders) | 1/6 (2) | 4/56 (7)
Localised oedema (General disorders) | 1/6 (2) | 0/56 (0)
Alanine amiontransferase increased (Investigations) | 6/6 (26) | 44/56 (155)
Haemoglobin decreased (Investigations) | 6/6 (23) | 42/56 (130)
White blood cell count decreased (Investigations) | 5/6 (40) | 52/56 (370)
Aspartate aminotransferase increased (Investigations) | 4/6 (24) | 38/56 (133)
Lymphocyte count decreased (Investigations) | 4/6 (22) | 28/56 (101)
Neutrophil count decreased (Investigations) | 4/6 (39) | 54/56 (368)
Platelet count decreased (Investigations) | 4/6 (22) | 39/56 (164)
Blood alkaline phosphatase increased (Investigations) | 4/6 (7) | 14/56 (23)
Red blood cell count decreased (Investigations) | 3/6 (8) | 37/56 (112)
Platelet count increased (Investigations) | 3/6 (17) | 10/56 (33)
Gamma-glutamyltransferase increased (Investigations) | 2/6 (3) | 18/56 (23)
Glucose urine present (Investigations) | 2/6 (2) | 4/56 (11)
Haematocrit decreased (Investigations) | 2/6 (11) | 32/56 (116)
Blood urine present (Investigations) | 2/6 (3) | 8/56 (13)
Weight decreased (Investigations) | 2/6 (3) | 3/56 (3)
Protein urine present (Investigations) | 2/6 (5) | 8/56 (15)
Blood albumin decreased (Investigations) | 1/6 (4) | 13/56 (25)
Blood bilirubin increased (Investigations) | 1/6 (1) | 6/56 (10)
Blood calcium decreased (Investigations) | 1/6 (4) | 2/56 (2)
Blood calcium increased (Investigations) | 1/6 (2) | 2/56 (6)
Blood pressure increased (Investigations) | 1/6 (1) | 4/56 (14)
Blood sodium decreased (Investigations) | 1/6 (1) | 5/56 (9)
Leucine aminopeptidase increased (Investigations) | 1/6 (1) | 0/56 (0)
Neutrophil count increased (Investigations) | 1/6 (1) | 7/56 (10)
Weight increased (Investigations) | 1/6 (1) | 1/56 (1)
White blood cell count increased (Investigations) | 1/6 (1) | 7/56 (13)
Joint sprain (Injury, poisoning and procedural complications) | 1/6 (1) | 0/56 (0)
Cautery to nose (Surgical and medical procedures) | 1/6 (2) | 0/56 (0)
Cellulitis (Infections and infestations) | 0/6 (0) | 3/56 (3)
Hordeolum (Infections and infestations) | 0/6 (0) | 2/56 (2)
Gastroenteritis (Infections and infestations) | 0/6 (0) | 1/56 (1)
Genital herpes (Infections and infestations) | 0/6 (0) | 1/56 (1)
Infection (Infections and infestations) | 0/6 (0) | 1/56 (1)
Pulpitis dental (Infections and infestations) | 0/6 (0) | 1/56 (1)
Lentigo (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/6 (0) | 1/56 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/6 (0) | 1/56 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0/6 (0) | 2/56 (2)
Seasonal allergy (Immune system disorders) | 0/6 (0) | 1/56 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0/6 (0) | 1/56 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0/6 (0) | 1/56 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0/6 (0) | 1/56 (1)
Agitation (Psychiatric disorders) | 0/6 (0) | 1/56 (1)
Anxiety (Psychiatric disorders) | 0/6 (0) | 1/56 (1)
Hyperaesthesia (Nervous system disorders) | 0/6 (0) | 2/56 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0/6 (0) | 2/56 (2)
Dizziness postural (Nervous system disorders) | 0/6 (0) | 1/56 (1)
Neuralgia (Nervous system disorders) | 0/6 (0) | 1/56 (1)
Neurotoxicity (Nervous system disorders) | 0/6 (0) | 1/56 (6)
Parosmia (Nervous system disorders) | 0/6 (0) | 1/56 (1)
Sciatica (Nervous system disorders) | 0/6 (0) | 1/56 (1)
Somnolence (Nervous system disorders) | 0/6 (0) | 1/56 (7)
Syncope vasovagal (Nervous system disorders) | 0/6 (0) | 1/56 (1)
Vocal cord paralysis (Nervous system disorders) | 0/6 (0) | 1/56 (1)
Olfactory nerve disorder (Nervous system disorders) | 0/6 (0) | 1/56 (4)
Eye discharge (Eye disorders) | 0/6 (0) | 3/56 (3)
Ocular hyperaemia (Eye disorders) | 0/6 (0) | 3/56 (3)
Conjunctival haemorrhage (Eye disorders) | 0/6 (0) | 1/56 (1)
Diplopia (Eye disorders) | 0/6 (0) | 1/56 (1)
Eyelid oedema (Eye disorders) | 0/6 (0) | 1/56 (2)
Lacrimation increased (Eye disorders) | 0/6 (0) | 1/56 (1)
Vision blurred (Eye disorders) | 0/6 (0) | 1/56 (1)
Tinnitus (Ear and labyrinth disorders) | 0/6 (0) | 1/56 (1)
Vertigo (Ear and labyrinth disorders) | 0/6 (0) | 1/56 (1)
Arrhythmia (Cardiac disorders) | 0/6 (0) | 1/56 (1)
Atrial fibrillation (Cardiac disorders) | 0/6 (0) | 1/56 (1)
Tachycardia (Cardiac disorders) | 0/6 (0) | 1/56 (1)
Ventricular extrasystoles (Cardiac disorders) | 0/6 (0) | 1/56 (1)
Hot flush (Vascular disorders) | 0/6 (0) | 6/56 (13)
Vasculitis (Vascular disorders) | 0/6 (0) | 3/56 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 9/56 (11)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 4/56 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 3/56 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 2/56 (3)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 2/56 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 1/56 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 1/56 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 1/56 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0/6 (0) | 1/56 (2)
Diarrhoea (Gastrointestinal disorders) | 0/6 (0) | 13/56 (27)
Stomach discomfort (Gastrointestinal disorders) | 0/6 (0) | 5/56 (8)
Abdominal distension (Gastrointestinal disorders) | 0/6 (0) | 4/56 (4)
Abdominal pain (Gastrointestinal disorders) | 0/6 (0) | 3/56 (5)
Cheilitis (Gastrointestinal disorders) | 0/6 (0) | 3/56 (3)
Haemorrhoids (Gastrointestinal disorders) | 0/6 (0) | 3/56 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0/6 (0) | 2/56 (3)
Dyspepsia (Gastrointestinal disorders) | 0/6 (0) | 2/56 (5)
Gastritis (Gastrointestinal disorders) | 0/6 (0) | 2/56 (2)
Stomatitis (Gastrointestinal disorders) | 0/6 (0) | 2/56 (4)
Gingival bleeding (Gastrointestinal disorders) | 0/6 (0) | 1/56 (5)
Gingival pain (Gastrointestinal disorders) | 0/6 (0) | 1/56 (1)
Gingival swelling (Gastrointestinal disorders) | 0/6 (0) | 1/56 (1)
Gingivitis (Gastrointestinal disorders) | 0/6 (0) | 1/56 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0/6 (0) | 1/56 (1)
Rash (Skin and subcutaneous tissue disorders) | 0/6 (0) | 16/56 (26)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0/6 (0) | 4/56 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0/6 (0) | 2/56 (5)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0/6 (0) | 2/56 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0/6 (0) | 2/56 (3)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0/6 (0) | 2/56 (2)
Blister (Skin and subcutaneous tissue disorders) | 0/6 (0) | 1/56 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0/6 (0) | 1/56 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0/6 (0) | 1/56 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 0/6 (0) | 1/56 (2)
Skin erosion (Skin and subcutaneous tissue disorders) | 0/6 (0) | 1/56 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0/6 (0) | 1/56 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 4/56 (8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 3/56 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 3/56 (4)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 2/56 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 1/56 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 1/56 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 1/56 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0/6 (0) | 1/56 (1)
Residual urine (Renal and urinary disorders) | 0/6 (0) | 3/56 (3)
Dysuria (Renal and urinary disorders) | 0/6 (0) | 1/56 (2)
Cystitis-like symptom (Renal and urinary disorders) | 0/6 (0) | 1/56 (2)
Breast discharge (Reproductive system and breast disorders) | 0/6 (0) | 1/56 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/6 (0) | 1/56 (1)
Fatigue (General disorders) | 0/6 (0) | 7/56 (15)
Face oedema (General disorders) | 0/6 (0) | 5/56 (9)
Pain (General disorders) | 0/6 (0) | 5/56 (8)
Chest discomfort (General disorders) | 0/6 (0) | 4/56 (4)
Oedema (General disorders) | 0/6 (0) | 3/56 (3)
Thirst (General disorders) | 0/6 (0) | 2/56 (2)
Asthenia (General disorders) | 0/6 (0) | 1/56 (1)
Chest pain (General disorders) | 0/6 (0) | 1/56 (1)
Feeling abnormal (General disorders) | 0/6 (0) | 1/56 (1)
Feeling drunk (General disorders) | 0/6 (0) | 1/56 (1)
Generalised oedema (General disorders) | 0/6 (0) | 1/56 (1)
Hangover (General disorders) | 0/6 (0) | 1/56 (1)
Injection site reaction (General disorders) | 0/6 (0) | 1/56 (1)
Local swelling (General disorders) | 0/6 (0) | 1/56 (1)
Blood potassium decreased (Investigations) | 0/6 (0) | 10/56 (23)
Protein total decreased (Investigations) | 0/6 (0) | 9/56 (21)
Blood lactate dehydrogenase increased (Investigations) | 0/6 (0) | 7/56 (24)
Blood creatinine increased (Investigations) | 0/6 (0) | 6/56 (7)
Blood urea decreased (Investigations) | 0/6 (0) | 6/56 (10)
C-reactive protein increased (Investigations) | 0/6 (0) | 4/56 (8)
Blood chloride decreased (Investigations) | 0/6 (0) | 3/56 (4)
Blood triglycerides increased (Investigations) | 0/6 (0) | 3/56 (6)
White blood cells urine positive (Investigations) | 0/6 (0) | 3/56 (3)
Blood cholesterol increased (Investigations) | 0/6 (0) | 2/56 (7)
Blood glucose increased (Investigations) | 0/6 (0) | 2/56 (7)
Blood potassium increased (Investigations) | 0/6 (0) | 2/56 (2)
Blood urea increased (Investigations) | 0/6 (0) | 2/56 (2)
Creatine phosphokinase decreased (Investigations) | 0/6 (0) | 2/56 (4)
Alanine aminotransferase decreased (Investigations) | 0/6 (0) | 1/56 (1)
Aspartate aminotransferase decreased (Investigations) | 0/6 (0) | 1/56 (2)
Blood cholinesterase increased (Investigations) | 0/6 (0) | 1/56 (1)
Blood creatinine decreased (Investigations) | 0/6 (0) | 1/56 (1)
Blood pressure decreased (Investigations) | 0/6 (0) | 1/56 (1)
Blood sodium increased (Investigations) | 0/6 (0) | 1/56 (2)
Glycosylated haemoglobin increased (Investigations) | 0/6 (0) | 1/56 (1)
Haematocrit increased (Investigations) | 0/6 (0) | 1/56 (1)
High density lipoprotein increased (Investigations) | 0/6 (0) | 1/56 (2)
Low density lipoprotein increased (Investigations) | 0/6 (0) | 1/56 (2)
Lymphocyte count increased (Investigations) | 0/6 (0) | 1/56 (3)
Urobilin urine present (Investigations) | 0/6 (0) | 1/56 (2)
Contusion (Injury, poisoning and procedural complications) | 0/6 (0) | 2/56 (3)
Wound (Injury, poisoning and procedural complications) | 0/6 (0) | 2/56 (2)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0/6 (0) | 1/56 (3)
Animal bite (Injury, poisoning and procedural complications) | 0/6 (0) | 1/56 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0/6 (0) | 1/56 (1)
Head injury (Injury, poisoning and procedural complications) | 0/6 (0) | 1/56 (1)
Central venous catheterisation (Surgical and medical procedures) | 0/6 (0) | 4/56 (4)
Catheterisation venous (Surgical and medical procedures) | 0/6 (0) | 1/56 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days